CLINICAL TRIAL: NCT00755690
Title: Study of Dietary Phosphate and Mineral Homeostasis in Early Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H08-01018
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Kidney Diseases
Keywords: Chronic Kidney Disease; CKD; Diet; Dietary Phosphate; Mineral Metabolism; FGF-23
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): High/ Low Phosphate diet I. A five-day low phosphate diet / A five-day low phosphate diet with the addition of a phosphate binder / A five-day high phosphate diet.
  II. A five-day low phosphate diet / A five-day high phosphate diet / A five-day low phosphate diet with the addition of a phosphate binder III. A five-day high phosphate diet / A five-day low phosphate diet with the addition of a phosphate binder / A five-day low phosphate diet.
  IV. A five-day high phosphate diet / A five-day low phosphate diet / A five-day low phosphate diet with the addition of a phosphate binder.
  V. A five-day low phosphate diet with the addition of a phosphate binder / A five-day low phosphate diet / A five-day high phosphate diet.
  VI. A five-day low phosphate diet with the addition of a phosphate binder / A five-day high phosphate diet / A five-day low phosphate diet.
  Interventions: Behavioral: High/ Low Phosphate diet
- 2 (Active Comparator): High/ Low Phosphate diet
  Interventions: Behavioral: High/ Low Phosphate diet
- 3 (Active Comparator): High/ Low Phosphate diet
  Interventions: Behavioral: High/ Low Phosphate diet

INTERVENTIONS:
Behavioral: High/ Low Phosphate diet — Low phosphate diet (750mg/day).
  Arms: 1
Behavioral: High/ Low Phosphate diet — Low phosphate diet (750mg/day) with the addition of the phosphate binder aluminum hydroxide (500mg three times per day).
  Arms: 2
Behavioral: High/ Low Phosphate diet — III. High phosphate diet (2000mg /day).
  Arms: 3

SUMMARY:
This study is designed to describe the physiological response to increased and decreased dietary phosphate intake on various parameters of mineral metabolism in the blood and urine of individuals with Chronic Kidney Disease stage 3 and 4 with normal serum phosphate levels. This detailed study will give us a far greater understanding of the role of diet in abnormal mineral homeostasis early in the progression of this chronic disease. The findings of this study will help both physicians and dietitians better determine the optimal time to introduce dietary therapy in CKD.

DETAILED DESCRIPTION:
The potential benefits of implementation of phosphate management earlier in CKD (Stages 3/4) are threefold: 1) prevention of vascular damage early in the progression of CKD thus reducing risk of cardiovascular death 2) Improved management of renal bone disease and resultant co-morbidities and 3) slowing the progression of renal failure lengthening the time required till dialysis is required. Although dietary counseling is currently a normal part of CKD care, the utility and effectiveness of lowering phosphate has not previously been quantified. In part this is due to the difficulty of measurement of serum phosphate as it is so tightly controlled before GFR falls below 30mls/min. No studies have investigated whether is it possible to modulate circulating FGF-23 and phosphate excretion in early stages of renal failure using diet in individuals with normal serum phosphate levels.

Study Objectives ;

1. To measure FGF-23 levels before and after a high phosphate diet, low phosphate diet and a low phosphate diet with phosphate binders.
2. To measure levels of calcium, phosphate, PTH, 25 and 1,25 vitamin D and fractional phosphate excretion before and after a high phosphate diet, low phosphate diet and a low phosphate diet with phosphate binders.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients with CKD stage 3 and 4 (eGFR < 60 ml/min and > 15 ml/min per 1.73 m2, not requiring dialysis).
* Normal serum phosphate stable over three months (> 0.87 mmol/L and < 1.70 mmol/L)
* Not yet following a low phosphate diet as reported by the patient or the renal dietitian (<1500mg/d)
* Over 19 years of age

Exclusion Criteria:

* Body mass index <20 kg/m2
* Current use of phosphate binders or active vitamin D or phenytonin (which induces vitamin D catabolism)
* Primary parathyroid defects
* Diagnosed osteoporosis
* Gut absorption defects
* Liver disease
* Pregnancy or lactation
* Patients hospitalised within the last 4 weeks

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
FGF-23 | 5 days

SECONDARY OUTCOMES:
Serum calcium, phosphate, PTH, 25 and 1,25 vitamin D and fractional phosphate excretion. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Adeera Levin, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada